CLINICAL TRIAL: NCT05273359
Title: Immunological Basis for Benralizumab Activity in Chronic Obstructive Pulmonary Disease (COPD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Temple University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ESR-19-20357
Record Dates: First submitted 2022-01-12; First posted 2022-03-10 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — benralizumab; Population Groups

STUDY DESIGN:
Intervention Model Description: A pilot double-blind randomized and placebo-controlled trial; participants will be blinded to the drug group; investigational pharmacist will be unblinded.
Who Masked: Participant
Masking Description: Placebo group: 15 subjects (>220 eosinophils/microliter) will receive a matching benralizumab placebo subcutaneous injection every 4 weeks for 4 complete doses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Benralizumab Intervention (Active Comparator): 15 subjects (≥220 eosinophils/microliter) will receive benralizumab 100 mg subcutaneous injection every 4 weeks for 4 complete doses.
  Interventions: Drug: Benralizumab
- Benralizumab Placebo (Placebo Comparator): 15 subjects (>220 eosinophils/microliter) will receive a matching benralizumab placebo subcutaneous injection every 4 weeks for 4 complete doses.
  Interventions: Other: Benralizumab placebo
- Comparison (control) group; no intervention (Other): 15 subjects (<150 eosinophils/microliter) will not receive any intervention.
  Interventions: Other: Comparison (control) group; no intervention

INTERVENTIONS:
Drug: Benralizumab — 15 subjects (≥220 eosinophils/microliter) will receive benralizumab 100 mg subcutaneous injection every 4 weeks for 4 complete doses.
  Arms: Benralizumab Intervention
Other: Benralizumab placebo — 15 subjects (>220 eosinophils/microliter) will receive a matching benralizumab placebo subcutaneous injection every 4 weeks for 4 complete doses.
  Arms: Benralizumab Placebo
Other: Comparison (control) group; no intervention — 15 subjects (<150 eosinophils/microliter) will not receive any intervention.
  Arms: Comparison (control) group; no intervention

SUMMARY:
The current literature suggests that the mode of action of benralizumab is to deplete eosinophils through a mechanism of antibody-dependent cell-mediated cytotoxicity. This direct cellular cytotoxicity may not explain all of the benralizumab effects. The investigators propose a set of studies to systematically examine the spectrum of effects of this drug on the immune system.

DETAILED DESCRIPTION:
The investigators will recruit a total of 45 Chronic Obstructive Pulmonary Disease (COPD) participants from the Temple University Hospital Lung Center Clinic. All participants will have moderate to severe COPD and have a history of 2 or more acute exacerbations in the past year. Thirty participants will have eosinophil counts of greater than 220 cells/microliter and 15 participants will have an eosinophil count less than 150 cells/microliter. The 15 participants with eosinophil counts less than 150 cells/microliter will be similar in age, gender, race, and disease burden to the 30 participants in the treatment arms. The investigators studies will include an analysis of the status of the systemic and lung inflammatory phenotype of the major leukocyte populations, using multiparameter flow cytometry. The investigators will couple these studies with an analysis of a panel of inflammatory and anti-inflammatory biomarkers in both the blood and bronchoalveolar lavage fluid. Very importantly, the investigators will characterize the functional capacity of T cells, B cells, monocytes, and granulocytes during drug therapy. These assessments will be linked to a characterization of the immunocompetence of the leukocytes by assessing global transcript dynamics as determined by RNA sequencing (RNAseq). Finally, the investigators will determine the influence of drug treatment by conducting metagenomic sequencing of bacterial, fungal and viral components of the microbiome in these patients. By using this approach, the investigators believe that a more complete understanding of the scope of activity of benralizumab at the level of immune competence will be developed.

ELIGIBILITY:
Inclusion Criteria:

Current smoker or ex-smoker with a tobacco history of ≥10 pack-years (1 pack year = 20 cigarettes smoked per day for 1 year). (Note: electronic cigarette [e-cigarette] use does not contribute to the pack-year count for eligibility).

History of moderate to very severe Chronic Obstructive Pulmonary Disease (COPD) with a post-bronchodilator forced expiratory volume in the first second (FEV1)/forced vital capacity (FVC) <0.70 and a post-bronchodilator FEV1 ≤ 65% of predicted normal value at screening central spirometry assessment.

Documented history of 2 or more moderate and/or severe COPD exacerbations in the past year that required treatment with systemic corticosteroids (at least 3 days or a single depot formulation injection) and/or hospitalization within 52 weeks prior to enrollment.

1. Exacerbations treated with antibiotics alone are not considered as meeting the criterion unless it is accompanied by treatment with systemic corticosteroids and/or hospitalization.
2. Hospitalization is defined as an inpatient admission ≥ 24 hours in the hospital, in an observation area, the emergency department, or other equivalent healthcare facility depending on the country and healthcare system.
3. Previous exacerbations should be confirmed to have occurred while patient was on stable triple Inhaled Corticosteroid (ICS)/ Long-Acting Beta2-Agonist (LABA)/ Long-Acting Muscarinic Antagonist (LAMA) background therapy for COPD and not as a result of a step down in therapy, i.e. change from triple to dual therapy.

Documented use of triple (ICS/LABA/LAMA) background therapy for COPD throughout the year (52 weeks) prior to enrollment.

1. ICS in a dose approved for COPD or equivalent or greater than 250 mcg of fluticasone propionate daily.
2. Patient could have switched therapies during the previous year and/or stepped down for short periods of time, although the total cumulative duration that the patient was not using triple (ICS/LABA/LAMA) background therapy must not exceed 2 months.
3. Patient must be on stable therapy/doses for the last 3 months prior to randomization. (Individual component changes or switches between devices are allowed as long as the patient remains on ICS/LABA/LAMA with an acceptable ICS dose).

For the 30 patients that will be randomized to treatment, blood eosinophil counts must be ≥ 220 cells/μL at screening (Temple Hospital lab), supported by at least 1 documented historical blood eosinophil count of ≥150 cells/microliter within 52 weeks of enrollment. In the absence of historical data, an additional blood eosinophil count must be obtained by repeating the testing during the run-in period (at least 4 weeks apart) with a result of >=220 cells/microliter. For the 15 patients in the comparison group, blood eosinophil count <150 cells/microliter at screening central laboratory testing. In the absence of historical data, an additional blood eosinophil count must be obtained by repeating the testing during the run-in period (at least 4 weeks apart) with a result of <150 cells/microliter.

COPD assessment test (CAT) total score ≥ 15 at Visit 1. Ability to read and write English.

Reproduction Negative pregnancy test (serum) for female patients of childbearing potential at Visit 1 (enrollment).

Women of childbearing potential (WOCBP) must agree to use a highly effective method of birth control (confirmed by the investigator) from enrollment throughout the study duration and within 12 weeks after last dose of IP. Highly effective forms of birth control include:

* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation- oral, intravaginal, or transdermal
* Progestogen-only hormonal contraception associated with inhibition of ovulation- oral, injectable, or implantable
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Sexual abstinence, i.e. refraining from heterosexual intercourse (The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical study and the preferred and usual lifestyle of the patient.)
* Vasectomized sexual partner (provided that partner is the sole sexual partner of the WOCBP study patient and that the vasectomized partner has received medical assessment of the surgical success) In addition to agreeing to use a highly effective form of birth control, WOCBP will be counseled at each visit regarding the importance of practicing birth control during the course of the study and not becoming pregnant. Urine pregnancy testing will be performed and a negative pregnancy test documented at each clinic visit.

Women not of childbearing potential are defined as women who are either permanently sterilized (hysterectomy, bilateral oophorectomy, or bilateral salpingectomy), or who are postmenopausal. Women will be considered postmenopausal if the woman has been amenorrheic for ≥12 months prior to the planned date of randomization without an alternative medical cause. The following age-specific requirements apply:

* Women <50 years old will be considered postmenopausal if the woman has have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatment and follicle stimulating hormone (FSH) levels in the postmenopausal range.
* Women ≥50 years old will be considered postmenopausal if the woman has been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatment.

Exclusion Criteria:

1. Clinically important pulmonary disease other than COPD (e.g. active lung infection, clinically significant bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia).
2. Current diagnosis of asthma according to the Global Initiative for Asthma (GINA) or other accepted guidelines, prior history of asthma, or asthma-COPD overlap according to GINA/Global Initiative for Obstructive Lung Disease (GOLD). Childhood history of asthma is allowed and defined as asthma diagnosed and resolved (i.e. not requiring use of any maintenance or rescue medication) before the age of 18.
3. Radiological findings suggestive of a respiratory disease other than COPD that is contributing to the patient's respiratory symptoms. Radiological findings of a solitary pulmonary nodule without appropriate follow up and demonstration of stability as per standard of care or findings suggestive of acute infection.
4. Another diagnosed pulmonary or systemic disease that is associated with elevated peripheral eosinophil counts (e.g. allergic bronchopulmonary aspergillosis/mycosis, eosinophilic granulomatosis with polyangiitis, hypereosinophilic syndrome).
5. Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the investigator and/or could:

   * Affect the safety of the patient throughout the study
   * Influence the findings of the study or their interpretation
   * Impede the patient's ability to complete the entire duration of the study
6. Signs and/or symptoms of cor pulmonale and/or right ventricular failure.
7. Patients receiving long-term oxygen treatment >4.0 liters/minute (L/min). While breathing supplemental oxygen, patients should demonstrate an oxyhemoglobin saturation ≥ 89%. In order to be admitted to the study, patients on long-term oxygen therapy have to be ambulatory and be able to attend clinic visits.
8. Use, or need for chronic use, of any non-invasive positive pressure ventilation device (NIPPV). Note: Patients using continuous positive airway pressure (CPAP) for Sleep Apnea Syndrome are allowed in the study.
9. History of known immunodeficiency disorder including a positive test for human immunodeficiency virus, HIV-1 or HIV-2.
10. Active liver disease. Chronic stable hepatitis B and C (including positive testing for hepatitis B surface antigen or hepatitis C antibody), or other stable chronic liver disease are acceptable if patient otherwise meets eligibility criteria. Stable chronic liver disease is defined by the absence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, or persistent jaundice, or cirrhosis.
11. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) level ≥ 3 times the upper limit of normal (ULN), confirmed by repeated testing during the run-in period. Transient increase of AST/ALT level that resolves by the time of randomization is acceptable if, in the investigator's opinion, the patient does not have an active liver disease and meets other eligibility criteria.
12. A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.
13. History of alcohol or drug abuse within the past year, which may compromise the study data interpretation as judged by investigator.
14. Malignancy, current or within the past 5 years, except for adequately treated non-invasive basal cell and squamous cell carcinoma of the skin or cervical carcinoma-in-situ treated with apparent success more than 1 year prior to Visit 1. Suspected malignancy or undefined neoplasms.
15. Patients who, in the opinion of the investigator or qualified designee, have evidence of active Tuberculosis (TB). Patients with a recent (within 2 years) first-time or newly positive purified protein derivative (PPD) test or Quantiferon test need to complete an appropriate course of treatment before being considered for enrollment. Evaluation will be according to the local standard of care and may consist of history and physical examinations, chest X-ray, and/or TB test as determined by local guidelines.
16. Patients participating in, or scheduled for, an intensive (active) COPD rehabilitation program (patients who are in the maintenance phase of a rehabilitation program are eligible to take part).
17. Patients with a history of surgical or endoscopic (e.g. valves) lung volume reduction within the 6 months prior to enrollment. Patients with a history of partial or total lung resection (single lobe or segmentectomy is acceptable).
18. Scheduled major surgical procedure during the course of the study. Minor elective procedures are allowed.
19. History of anaphylaxis to benralizumab or any other biologic therapy. Prior/concomitant therapy
20. Receipt of blood products or immunoglobulins within 30 days prior to randomization.
21. Receipt of any marketed or investigational biologic product for any reason within 4 months or 5 half-lives prior to randomization, whichever is longer.
22. Receipt of live attenuated vaccines 30 days prior to randomization.
23. Chronic use of immunosuppressive medication (including but not limited to: methotrexate, troleandomycin, cyclosporine, azathioprine, rectal corticosteroids, and systemic corticosteroids) or expected need for chronic use during the study.
24. Chronic use of antibiotics if duration of treatment is <9 months prior to randomization (Visit 3). Chronic macrolide or other antibiotic therapy is allowed provided the patient has been on a stable dose/regimen for ≥ 9 months prior to randomization and has had ≥ 2 COPD exacerbations in the past year while on stable therapy. If the patient was previously on chronic antibiotic but is no longer taking it, the patient cannot be randomized until 6 weeks after the last dose.

    Prior/concurrent clinical study experience
25. Receipt of any investigational non-biologic product within 30 days or 5 half-lives prior to enrollment, whichever is longer.
26. Receipt of benralizumab within 12 months prior to enrollment.
27. Known history of allergy or reaction to any component of the intraperitoneal (IP) formulation.

    Other exclusions
28. Donation of blood, plasma, or platelets within the past 90 days prior to enrollment.
29. Pregnant, breastfeeding, or lactating women.
30. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
31. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Lifestyle restrictions Women of childbearing potential must use highly effective contraceptive methods from enrollment throughout the study and for at least 12 weeks (≥ 5 half-lives) after last administration of the IP, as stated in inclusion criterion 11.

Patients must abstain from donating blood, plasma, or platelets from the time of informed consent and for 12 weeks (≥ 5 half-lives) after last dose of IP.

-

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline of peripheral blood eosinophil and B cell levels | The duration of a subject's participation in the research study is 6 months for those patients with eosinophil counts ≥220 cells/microliter and 1 day for those patients with eosinophil counts <150 cells/microliter.
  Peripheral blood eosinophil and B cell number counts

SECONDARY OUTCOMES:
Change from baseline of peripheral blood T cells | 6 months
  Peripheral blood T cell number counts
Change from baseline of peripheral blood monocytes | 6 months
  Peripheral blood monocyte number counts
Change from baseline of peripheral blood neutrophils | 6 months
  Peripheral blood neutrophil cell number counts
Change from baseline of peripheral blood NK cells | 6 months
  Peripheral blood NK cell number counts
Change from baseline of peripheral blood dendritic cells | 6 months
  Peripheral blood dendritic cell number counts
Change from baseline of peripheral blood IL-4 levels | 6 months
  Blood IL-4 pg/ml
Change from baseline of peripheral blood IL-5 levels | 6 months
  Blood IL-5 pg/ml
Change from baseline of peripheral blood IL-13 levels | 6 months
  Blood IL-13 pg/ml
Change from baseline of peripheral blood CCL24 levels | 6 months
  Blood CCL24 pg/ml
Change from baseline of peripheral blood CCL26 levels | 6 months
  Blood CCL26 pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rogers, PhD, Principal Investigator — Temple University